CLINICAL TRIAL: NCT00531011
Title: EXecutive Randomized Controlled Trial (RCT): XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS) in the Treatment of the Specific Setting of Patients With Multi-vessel Coronary Artery Disease.
Brief Title: EXecutive RCT: Evaluating XIENCE V® in a Multi Vessel Disease
Acronym: EXecutive
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-380 RCT
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Artery Stenosis; Coronary Artery Restenosis
Keywords: Stents; Drug-eluting Stent; Angioplasty; Coronary Artery stenosis; Coronary Artery Stent Restenosis; Stent Thrombosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XIENCE V (Active Comparator): Patients randomized to receive the XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS)
  Interventions: Device: XIENCE V® Everolimus Eluting Coronary Stent System
- TAXUS® Liberté™ (Active Comparator): Patients randomized to receive the TAXUS® Liberté™ Paclitaxel Eluting Coronary Stent System
  Interventions: Device: TAXUS® Liberté™ Paclitaxel Eluting Coronary Stent System

INTERVENTIONS:
Device: XIENCE V® Everolimus Eluting Coronary Stent System — Coronary artery placement of a drug-eluting stent
  Arms: XIENCE V
Device: TAXUS® Liberté™ Paclitaxel Eluting Coronary Stent System — Coronary artery placement of a drug-eluting stent
  Arms: TAXUS® Liberté™

SUMMARY:
The purpose of this two part study is the assessment of the performance of the XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS) in the treatment of the specific setting of patients with Multi-Vessel Coronary Artery Disease (MVD).

DETAILED DESCRIPTION:
This is a clinical evaluation of the XIENCE V® everolimus eluting coronary stent system as a revascularization treatment of patients with multi-vessel coronary artery disease (MVD-CAD).

The long term safety and efficacy of the XIENCE V EECSS have been demonstrated in the SPIRIT FIRST trial up to 5 years, the SPIRIT II trial up to 4 years, and in the SPIRIT III Randomized Control Trial (RCT) up to 3 years. In addition, these pre-approval studies have shown low rates of Target Vessel Failure and Major Adverse Cardiac Events (MACE) that were consistently lower than the comparator arm of each study.

The post approval EXECUTIVE study demonstrated that the use of the XIENCE EECSS in complex lesions in a real-world population resulted in 1 year MACE, Stent Thrombosis and Target Lesion Revascularization rates that are comparable to those of the previously mentioned pre-approval studies which included patients with more restricted inclusion / exclusion criteria.

Therefore, based on existing data from these trials, Abbott Vascular has decided to discontinue further follow up in the EXECUTIVE trial.

The study is composed of two parts:

A Registry, outlined in a separate posting and the Randomized Control Trial (RCT) portion of this study, which is as follows:

-A randomized group of patients aimed at assessing the angiographic efficacy of the XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS) compared to the TAXUS® Liberté™ Paclitaxel Eluting Coronary Stent System.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years of age
2. Patient is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the XIENCE V® EECSS and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure, as approved by the appropriate Medical Ethics Committee of the respective clinical site
3. Patient has been diagnosed a MVD, as documented by coronary angiography, i.e. presenting a severe stenosis (>50%) amenable to PCI in at least 2 major epicardial vessels or their principal bifurcation branches (diagonal or obtuse marginal)
4. Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible change in the electrocardiogram -ECG- consistent with ischemia)
5. Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery
6. Patient must agree to undergo all protocol-required follow-up examinations.

Angiographic Inclusion Criteria

1. Patients may receive up to 4 planned XIENCE V® EECSS stents, depending on the number of vessels treated and their respective lesion length. When multiple lesions are present in one or more main coronary branches, complete revascularization should be attempted with the implantation of a maximum of 4 planned stents
2. Target lesions must be de novo lesions (no prior stent implant, no prior brachytherapy)
3. Target vessel reference diameter must be between 2.5 mm and 4.0 mm by visual estimate
4. Target lesion < or = 28 mm in length by visual estimation
5. Target lesions must be in a major artery or its principal branches (diagonal or obtuse marginal) with a visually estimated stenosis of > or = 50%
6. Two lesions in a single main coronary artery or its branches do not constitute a MVD situation, therefore this type of patient must not be enrolled

Exclusion Criteria:

1. Patient has had a known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure (non-procedural/spontaneous MI, CK-MB > or = to 2 times upper limit of normal) and CK and CK-MB have not returned within normal limits at the time of procedure
2. Patient has current unstable arrhythmias
3. Patient has a known left ventricular ejection fraction (LVEF) <30%
4. Patient has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant
5. Patient is receiving or scheduled to receive chemotherapy or radiation therapy within 30 days prior to or after the procedure.
6. Patient is receiving immunosuppression therapy or has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.)
7. Patient is receiving chronic anticoagulation therapy (e.g. coumadin)
8. Patient has a known hypersensitivity or contraindication to aspirin, paclitaxel, either heparin or bivalirudin, clopidogrel or ticlopidine, everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated
9. Elective surgery is planned within the first 9 months (+/- 14 days) after the procedure that will require discontinuing either aspirin or clopidogrel
10. Patient has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3, a WBC of <3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis)
11. Patient has known renal insufficiency (e.g., serum creatinine level of more than 2.5 mg/dl, patient on dialysis)
12. Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
13. Patient has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
14. Patient has had a significant GI or urinary bleed within the past six months
15. Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e. less than one year)
16. Patient is already participating in another investigational use device or drug study or has completed the follow-up phase of another study within the last 30 days.

Angiographic Exclusion Criteria

1. Target lesion meets any of the following criteria:

   * Left main location
   * Located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft (defined as vessel irregularity per angiogram and >20% stenosed lesion by visual estimation)
   * Heavy calcification
2. The patient may need more than 4 planned stents. Bailout stents are allowed but must be of the same type as randomization stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Vassanelli, MD, Principal Investigator — Ospedale Civile Maggiore - Università di Verona; Flavio Ribichini, MD, Principal Investigator — Ospedale Civile Maggiore - Università di Verona
Locations (24):
- Italy (24):
  - A.O. San Giovanni di Dio, Agrigento
  - Ospedale Maggiore Bologna, Bologna
  - Policlinico S. Orsola - Malpighi, Bologna
  - A.O. Cannizzaro, Catania
  - A.O. Universitaria Vittorio Emanuele - Ferrarotto - S. Bambino, Catania
  - A.O. Università Mater Domini c/o Campus Università Magna Grecia, Catanzaro
  - A.O. Universitaria OO.RR Foggia, Foggia
  - E.O. Ospedali Galliera, Genova
  - A.O. Carlo Poma, Mantova
  - Centro Cardiologico Monzino, Milan
  - Ospedale Loreto Mare, Napoli
  - A. O. Sant'Andrea, Roma
  - Ospedale Generale Madre Vannini, Roma
  - Ospedale Sandro Pertini, Roma
  - A.S.O. Molinette San Giovanni Battista di Torino, Torino
  - Ospedale Maria Vittoria, Torino
  - P.O. San Giovanni Bosco, Torino
  - San Giovanni Battista - Ospedale Molinette, Torino
  - A.O. Universitaria - Ospedale Riuniti Umberto I - G.M. Lancisi - G. Salesi, Torrette Di Ancona
  - Ospedale Civile Maggiore - Università di Verona, Verona
  - Ospedale Civile, Vicenza
  - Ospedale Civile di Vigevano, Vigevano
  - A.O. Della Provincia di Pavia, Voghera
  - Policlinico San Marco, Zingonia

REFERENCES:
- [Derived] Ribichini F, Romano M, Rosiello R, La Vecchia L, Cabianca E, Caramanno G, Milazzo D, Loschiavo P, Rigattieri S, Musaro S, Pironi B, Fiscella A, Amico F, Indolfi C, Spaccarotella C, Bartorelli A, Trabattoni D, Della Rovere F, Rolandi A, Beqaraj F, Belli R, Sangiorgio P, Villani R, Berni A, Sheiban I, Lopera Quijada MJ, Cappi B, Ribaldi L, Vassanelli C; EXECUTIVE Trial Investigators. A clinical and angiographic study of the XIENCE V everolimus-eluting coronary stent system in the treatment of patients with multivessel coronary artery disease: the EXECUTIVE trial (EXecutive RCT: evaluating XIENCE V in a multi vessel disease). JACC Cardiovasc Interv. 2013 Oct;6(10):1012-22. doi: 10.1016/j.jcin.2013.05.016. Epub 2013 Sep 18. PMID 24055444
- [Derived] Ribichini F, Ansalone G, Bartorelli A, Beqaraj F, Berni A, Colangelo S, D'Amico M, Della Rovere F, Fiscella A, Gabrielli G, Indolfi C, La Vecchia L, Loschiavo P, Marinoni G, Marzocchi A, Milazzo D, Romano M, Sangiorgio P, Sheiban I, Tamburino C, Tuccillo B, Villani R, Cappi B, Quijada MJ, Vassanelli C; EXECUTIVE Trial Investigators. A clinical and angiographic study of the XIENCE V everolimus-eluting coronary stent system in the treatment of patients with multivessel coronary artery disease. Study design and rationale of the EXECUTIVE trial. J Cardiovasc Med (Hagerstown). 2010 Apr;11(4):299-309. doi: 10.2459/JCM.0b013e3283331e69. PMID 20090550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patient population was comprised of male and female patients derived from the general interventional cardiology population from 9 centers in Italy.
Period: Overall Study
Arm/Group | XIENCE V | TAXUS® Liberté™
Started | 103 | 97
Completed | 99 | 90
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XIENCE V | TAXUS® Liberté™ | Total
Number analyzed (Participants) | 103 | 97 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 48 | 94
  >=65 years | 57 | 49 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.1) | 63.8 (10.2) | 64.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 76 | 73 | 149
Region of Enrollment [Number; unit: participants]
  Italy | 103 | 97 | 200

OUTCOME MEASURES:

1. Secondary Outcome: In-stent Binary Restenosis Rate
Description: This measures the percentage of patients who have > 50% diameter stenosis of the assessed vessel, within the stent edges.
Time Frame: at 9 months
Population: ITT, 167 patients performed angiographic follow-up.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Lesions
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 90 | 77
Number analyzed (Lesions) | 225 | 194
percentage of participants | 5.8 | 3.6

2. Secondary Outcome: In-segment Binary Restenosis Rate
Description: This measures the percentage of patients who have > 50% diameter stenosis of the assessed vessel, within the stent edges
  In-segment is measured within the confines of the stent edges plus within 5 mm on either side of the stent.
Time Frame: at 9 months
Population: 167 patients performed angiographic follow-up.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Lesions
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 90 | 77
Number analyzed (Lesions) | 225 | 194
percentage of participants | 6.2 | 4.6

3. Secondary Outcome: In-segment Late Loss (LL)
Description: LL is defined as the difference between the post-procedure (immediately post placement of the stent) minimal lumen diameter (MLD) and the follow-up MLD (at 270 days). In segment LL is measured within the confines of the stent edges and within 5 mm of those edges.
Time Frame: at 9 months
Population: 167 patients performed angiographic follow-up. Descriptive statistics for this measure are based on one random lesion per patient.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: lesions
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 90 | 77
Number analyzed (lesions) | 225 | 194
millimeters | -0.100 (0.484) | 0.037 (0.421)

4. Secondary Outcome: Composite Rate of Cardiac Death, Myocardial Infarction (MI, Both Q-wave and Non Q-wave), and Ischemia-driven Target Lesion Revascularization (TLR) .
Description: This measure is a calculation of the percentage of participants who experience any of the components of this composite measure.
Time Frame: at 30 days
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 103 | 97
percentage of participants | 1 | 2.1

5. Secondary Outcome: Composite Rate of All Death, MI (Q-wave and Non Q-wave), and Target Vessel Revascularization (TVR).
Time Frame: at 30 days
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 103 | 97
percentage of participants | 1 | 2.1

6. Secondary Outcome: Lesion Success
Description: defined as attainment of < 30% residual in-stent stenosis (by visual assessment) using any percutaneous method.
Time Frame: at the time of PCI
Population: Intent to treat (ITT)
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Lesions
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 103 | 97
Number analyzed (Lesions) | 259 | 234
Percentage of participants | 99.2 | 99.6

7. Secondary Outcome: Procedural Success
Description: defined as: residual in-stent %DS of < 30% using a percutaneous method, without cardiac death, Q-wave MI, non Q-wave MI, or repeat revasc of the target during hospitalization.
Time Frame: at the time of PCI
Measure: Number; unit: percentage of participants
Units Other Than Participants: Lesions
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 103 | 97
Number analyzed (Lesions) | 259 | 234
percentage of participants | 98.1 | 97

8. Secondary Outcome: Device Success
Description: defined as achievement of a final residual in-stent diameter stenosis of < 30% (visual assessment) using the assigned device only.
Time Frame: at the time of PCI
Measure: Number; unit: percentage of participants
Units Other Than Participants: Lesions
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 103 | 97
Number analyzed (Lesions) | 256 | 224
percentage of participants | 97.7 | 98.2

9. Secondary Outcome: Adjudicated Stent Thrombosis.
Time Frame: at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 103 | 97
percentage of participants | 0 | 0

10. Secondary Outcome: Adjudicated Stent Thrombosis.
Time Frame: 9 months
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 103 | 97
percentage of participants | 0 | 0

11. Secondary Outcome: Revascularizations
Description: (TLR/TVR/any revascularization)both ischemia-driven and not ischemia-driven.
Time Frame: at 30 days
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 103 | 97
percentage of participants | 0 | 0

12. Secondary Outcome: Revascularizations
Description: (TLR/TVR/any revascularization)both ischemia-driven and not ischemia-driven.
Time Frame: 9 months
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 103 | 97
percentage of participants | 5.8 | 11.3

13. Secondary Outcome: Composite Endpoint of Cardiac Death, MI (Q-wave and Non Q-wave), and Ischemia-driven TLR .
Description: ITT
Time Frame: 9 months
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 103 | 97
percentage of participants | 4.9 | 7.2

14. Secondary Outcome: Composite Endpoint of All Death, MI (Q-wave and Non Q-wave), and TVR.
Time Frame: 9 months
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 103 | 97
percentage of participants | 6.8 | 12.4

15. Secondary Outcome: In-stent Minimum Lumen Diameter (MLD).
Time Frame: at 9 months.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Lesions
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 90 | 77
Number analyzed (Lesions) | 225 | 194
millimeters | 2.29 (0.64) | 2.17 (0.61)

16. Secondary Outcome: In-segment Minimum Lumen Diameter (MLD).
Time Frame: at 9 months.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Lesions
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 90 | 77
Number analyzed (Lesions) | 225 | 194
millimeters | 2.10 (0.57) | 2.04 (0.52)

17. Secondary Outcome: Proximal Minimum Lumen Diameter (MLD).
Description: Proximal refers to the immediate 5 mm outside of the proximal end of the stent.
Time Frame: at 9 months.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Lesions
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 90 | 77
Number analyzed (Lesions) | 225 | 194
millimeters | 2.67 (0.65) | 2.61 (0.62)

18. Secondary Outcome: Distal Minimum Lumen Diameter (MLD).
Description: Distal refers to the immediate 5 mm outside of the distal end of the stent.
Time Frame: at 9 months.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Lesions
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 90 | 77
Number analyzed (Lesions) | 225 | 194
millimeters | 2.28 (0.59) | 2.25 (0.57)

19. Primary Outcome: In-stent Late Loss (LL)
Description: Full Analysis Set (FAS). LL is defined as the difference between the post-procedure (immediately post placement of the stent) minimal lumen diameter (MLD) and the follow-up MLD (at 270 days). In stent is measured within the confines of the stent edges.
Time Frame: at 270 days
Population: Descriptive statistics for this measure are based on one random lesion per patient, 167 patients performed angiographic follow-up.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Lesions
Arm/Group | XIENCE V | TAXUS® Liberté™
Number analyzed (Participants) | 90 | 77
Number analyzed (Lesions) | 225 | 194
millimeters | 0.052 (0.513) | 0.238 (0.504)

ADVERSE EVENTS:
Time Frame: 9 months
Description: Only serious adverse events were collected in the conduct of this trial. "Other" adverse events were not collected.
Arm/Group | XIENCE V | TAXUS® Liberté™
Serious Adverse Events (participants affected / at risk) | 21/101 | 19/91
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XIENCE V (N=101) | TAXUS® Liberté™ (N=91)
Cardiac death (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 6 (6) | 6 (6)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Thrombosis in device (General disorders) | 1 (1) | 0 (0)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 6 (6) | 10 (11)
Medical device complication (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) — Events under Mechanical complication are plaque shifts. There is no exact code for this event in MedDRA
Procedural complications (General disorders) | 2 (2) | 0 (0) — Events in this code wer failure of the stent to cross the lesion and failure of the wire to cross the lesion. There are no exact codes for these events in MedDRA.
Arteriogram coronary (Investigations) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Ischaemia NOS (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publication of the aggregate data is subject to the prior agreement of all the various sites participating in the study. Publication of the clinical data collected during the Study, can be only after notifying the SPONSOR in advance in order to allow the SPONSOR to verify compliance with confidentiality obligations and intellectual property rights of the SPONSOR.